CLINICAL TRIAL: NCT02404909
Title: Does Inferior Vena Cava Collapsibility Correlate With Fluid Regimen and Outcome in Patients Undergoing Liver Resection?
Brief Title: Inferior Vena Cava Index in Patients Undergoing Liver Resection
Acronym: IVC
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, MD, PhD, FACS, University of Milan
Other Study IDs: IVCindex
Record Dates: First submitted 2015-03-21; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with liver tumors candidate to hepatectomy
  Interventions: Other: IVC diameters evaluation by intraoperative ultrasound

INTERVENTIONS:
Other: IVC diameters evaluation by intraoperative ultrasound — Out of consecutive patients who underwent hepatectomy for primary and secondary liver tumors, patients in whom IVC diameters were intraoperatively measured for clinical reasons were retrospectively selected and analyzed

SUMMARY:
The aim of this study was to evaluate whether IVC index measured intraoperatively was affected by fluid administration and could add any helpful information about the hemodynamics during hepatic resection. In addition, the investigators evaluated whether IVC index was somehow correlated with the risk of postoperative complication.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent hepatectomy for primary and secondary liver tumors

Exclusion Criteria:

Patients with tumoral thrombosis or full tumoral involvement/compression of IVC were excluded. Patients unresectable at laparotomy for any extra-hepatic or intrahepatic reason and patients previously submitted to hepatectomy were not included

Ages: 34 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent liver resection for primary and secondary liver disease
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
to investigate the influence of the liver resection on hemodynamic status in terms of hemodynamic indexes changes | 4 weeks